CLINICAL TRIAL: NCT04294758
Title: Estimation of the Difference Between the Temperature of the Peritoneal Microenvironment and the Central Body Temperature During Laparoscopic Surgery. Prospective Observational Study
Acronym: TEMP-19
Status: Completed | Type: Observational
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: Principal Investigator, Oscar Diaz-Cambronero, Anesthetist, Hospital Universitario La Fe
Other Study IDs: FPR-IIS -029-02 Ed. 02
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Laparoscopic Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Estimation of the difference between the temperature of the peritoneal microenvironment and the central body temperature during laparoscopic surgery. Prospective observational study.

DETAILED DESCRIPTION:
Prospective unblinded observational study to measure the difference between central and peritoneal temperature during laparoscopic surgery.

CO2 insufflation at the peritoneal level to generate the pneumoperitoneum necessary to perform laparoscopic surgery results in a decrease in peritoneal temperature greater than that generated at the central level (esophageal temperature).

The potential long-term advantages of maintaining normothermia at the peritoneal level during laparoscopic surgery may derive from the reversal of the harmful effects of hypothermia at the level of the peritoneal microenvironment since the regional hypoxia resulting from vasoconstriction and the inhibition of functionality cellular that can favor complications such as bleeding or suture dehiscence.

On the other hand, the immune system can be affected by regional hypothermia in several ways. First, postoperative vasoconstriction restricts metabolic heat to the central regions of the body and accelerates overheating, but can simultaneously reduce tissue perfusion by inhibiting oxidative destruction of neutrophils, which is the first line of defense against bacterial contamination. Second, hypothermia reduces systemic immunity and decreases macrophage motility. Third, hypothermia reduces the recovery capacity necessary for wound contamination.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Classification of the American Society of Anesthesiologists (ASA I-III).
* Patients who do not have cognitive deficits.
* Prior signed informed consent.

Exclusion Criteria:

* Pregnancy or breastfeeding.
* Refusal of the patient to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing laparoscopic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Estimation of the difference between peritoneal and central temperature during laparoscopic surgery. | Since the beginning until the end of the surgery
Assess the difference between peritoneal and central temperature during laparoscopic surgery is modified with the total amount of insufflated gas and / or the duration of surgery. | Since the beginning until the end of the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital la Fe, Valencia, Spain

REFERENCES:
- [Derived] Mazzinari G, Rovira L, Vila Montanes M, Garcia Gregorio N, Ayas Montero B, Alberola Estelles MJ, Flor B, Argente Navarro MP, Diaz-Cambronero O. Estimation of the difference between peritoneal microenvironment and core body temperature during laparoscopic surgery - a prospective observational study. Sci Rep. 2024 Sep 2;14(1):20408. doi: 10.1038/s41598-024-71611-z. PMID 39223302